CLINICAL TRIAL: NCT00632918
Title: A Retrospective Study of Effects of Heart Rates and Variability of Heart Rates on Image Quality of Dual-Source CT Coronary Angiography With Regard to Motion Artifact.
Brief Title: Effects of Heart Rates and Variability of Heart Rates on Image Quality of Dual-Source CT Coronary Angiography
Acronym: DSCT
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Wing-Keung Cheung M.D. / Visiting Staff of Department of Medical Imaging in Far Easten Memorial Hospital, Department of Medical Imaging in Far Eastern Memorial Hospital
Other Study IDs: 96064
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: CT; Coronary Angiography
Keywords: Image quality; Dual-source CT; Coronary angiography; Heart rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: None Retained — No biospecimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to investigate the effects of heart rates (including maximum heart rate, average heart rate and minimum heart rate) and variability of heart rate on image quality of DSCT coronary angiography without control of heart rate experienced in our department.

DETAILED DESCRIPTION:
The dual-source CT (DSCT) equipped with two X-ray tubes at 90 degree offset in the gantry can provide temporal resolution 83ms using mono-segmental reconstruction technique. The recent studies about the effect of heart rate on IQ of DSCT coronary angiography which concluded in adequate diagnostic IQ of dual-source CTCA without immediate pre-scanning heart rate control included chronic users of β-blocker focused on the influences of average heart rate, heart rate variability and coronary arterial calcifications on IQ. The effect of blooming artifact of calcification on IQ by far cannot be eliminated. Here, we investigate the effects of maximum heart rate, average heart rate, minimum heart rate and heart rate variability on the motion-related IQ of DSCT coronary angiography in patients without both pre-scanning heart rate control and chronic use of β-blocker agent, compared with that in chronic users of β-blocker agents.

ELIGIBILITY:
Inclusion Criteria:

* From Oct 2006 to Jan 2007, CT coronary angiographies of 180 consecutive adult patients, were performed in our hospital using a DSCT scanner. After exclusion of the patients according to the exclusion criteria, totally DSCT coronary angiographies of 133 adult patients (N=133) were enrolled in this study. Among those 133 patients, including 97 males and 36 females with a mean age of 53.9 (ranging from 21 to 78 year old), 50 patients were chronic β-blocker users (group 1) while the other 83 patients (group 2) were not chronic user of any medication controlling heart rate

Exclusion Criteria:

* The patients below 18 year old, patients with status post heterotopic heart transplantation (having two hearts in a chest), patients with status post coronary by-pass surgery and patients with post indwelling of coronary arterial stents

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients or examined persons from Taiwan.
Sampling Method: Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2007-10; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Compare the effects of the heart rate variables on motion-related image qualities of DSCT coronary angiography between the group 1 patients of chronic beta-blocker users and the group 2 patients without medication of any heart-rate lowering agent. | About two months

SECONDARY OUTCOMES:
Kappa Statistics, Descriptive Statistics, Chi-square test, Independent t-test, Pearson's correlation and linear regression method for statistic analysis. | About two to three months

CONTACTS AND LOCATIONS:
Overall Officials: Wing-Keung Cheung, MD, CCD, Principal Investigator — Far Eastern Memorial Hospital; Kao-Lun Wang, MD, Study Chair — Far Eastern Memorial Hospital; Chen-I Yen, BSc, Study Chair — Far Eastern Memorial Hospital; Shu-Lin Tsen, BSc, Study Chair — Far Eastern Memorial Hospital
Locations (1):
- Department of Medical Imaing, Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan

REFERENCES:
- [Background] Leschka S, Scheffel H, Desbiolles L, Plass A, Gaemperli O, Valenta I, Husmann L, Flohr TG, Genoni M, Marincek B, Kaufmann PA, Alkadhi H. Image quality and reconstruction intervals of dual-source CT coronary angiography: recommendations for ECG-pulsing windowing. Invest Radiol. 2007 Aug;42(8):543-9. doi: 10.1097/RLI.0b013e31803b93cf. PMID 17620936
- [Background] Achenbach S, Ropers D, Kuettner A, Flohr T, Ohnesorge B, Bruder H, Theessen H, Karakaya M, Daniel WG, Bautz W, Kalender WA, Anders K. Contrast-enhanced coronary artery visualization by dual-source computed tomography--initial experience. Eur J Radiol. 2006 Mar;57(3):331-5. doi: 10.1016/j.ejrad.2005.12.017. Epub 2006 Jan 19. PMID 16426789
- [Result] Johnson TR, Nikolaou K, Wintersperger BJ, Leber AW, von Ziegler F, Rist C, Buhmann S, Knez A, Reiser MF, Becker CR. Dual-source CT cardiac imaging: initial experience. Eur Radiol. 2006 Jul;16(7):1409-15. doi: 10.1007/s00330-006-0298-y. Epub 2006 May 13. PMID 16770652
- [Result] Matt D, Scheffel H, Leschka S, Flohr TG, Marincek B, Kaufmann PA, Alkadhi H. Dual-source CT coronary angiography: image quality, mean heart rate, and heart rate variability. AJR Am J Roentgenol. 2007 Sep;189(3):567-73. doi: 10.2214/AJR.07.2078. PMID 17715102